CLINICAL TRIAL: NCT03999853
Title: Colonic Delivery of Butyrate to Improve Insulin Sensitivity and Lower Triglycerides in Type 1 Diabetes Subjects
Brief Title: Butyrate Adjuvant Therapy for Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: BioKier Inc. (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Adrian Vella, Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-006035
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Type1diabetes
Keywords: Butyrate
MeSH Terms: interventions — Butyrates

STUDY DESIGN:
Intervention Model Description: BKR-017: Delayed release butyrate which promotes endogenous incretin secretion to determine if this improves insulin action
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Conventional Therapy / Butyrate (Experimental): Subjects will be receiving usual therapy for the first study period (approx 1 month) then 500 mg Butyrate tablets to be taken at a dose of 1.5 g (3 tablets) twice daily (BID) for approx 2 months
  Interventions: Drug: BKR-017

INTERVENTIONS:
Drug: BKR-017 — BKR-017
  Other Names: Butyrate tablets

SUMMARY:
The investigators are interested to evaluate the effect of BKR-017 (colon-targeted 500 mg butyrate tablets) as adjuvant therapy on metabolic control in type 1 diabetes (TID) subjects.

DETAILED DESCRIPTION:
This study will test effect of BKR-017 (colon-targeted 500 mg butyrate tablets) as adjuvant therapy in type 1 diabetes (TID) Subjects on metabolic control in this population. Insulin sensitivity, glucose control (variability) and triglycerides will be measured after 8 weeks of treatment and compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

1. All type 1 diabetes with C-Peptide (CPR) less than 0.5 ng/mL subjects who are > 20 and <80 years of age recruited from the Mayo Clinic Endocrinology Clinic;
2. Will also meet HbA1c level of 6.4-8.9% and BMI of < 30 kg/m2 at week -4.

Exclusion Criteria:

1. Except for the use of insulin, no other treatments for T1D will be permitted.
2. Pregnancy
3. Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | (Day 0) to Day 28 and Day 56
  Change in Insulin sensitivity

SECONDARY OUTCOMES:
Glucose Variability and Triglycerides | (Day 0) to Day 28 and Day 56
  Changes in glucose measurements and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials